CLINICAL TRIAL: NCT00202956
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effects on Biomarkers and Safety of Bugusan (BGS) in Postmenopausal Patients With Osteoporosis.
Brief Title: Safety and Efficacy Study of Bugusan (BGS)to Treat Osteoporosis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JL-HM-01-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: Bugusan

SUMMARY:
The objective is to evaluate the effects on biomarkers and safety of BGS in postmenopausal patients with osteoporosis.

DETAILED DESCRIPTION:
The objective is to evaluate the effects on biomarkers and safety of BGS in postmenopausal patients with osteoporosis by a study of Randomized, Double Blind, Placebo-Controlled, Parallel Group.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women between the ages of 45 and 75 years with a natural menopause ≧ 6 months and serum E2 values < 20 pg/ml, serum FSH values ≧ 25 mIU/mL;
2. Patients have bone mineral density <-2.5 SD of T score at the lumbar spine (L2-L4);
3. All patients must sign the informed consent form (ICF) prior to the trial.

Exclusion Criteria:

1. Any X-ray film that documents substantial scoliosis, or spinal secondary osteoporosis;
2. Any X-ray film that documents bone fracture within 3 month prior to the trial.
3. Medication such as estrogen, bisphosphonates, calcitonin, fluoride, glucocorticoids, ipriflavone intake within 3 weeks prior to the trial;
4. Use of other Chinese medicine within 2 weeks prior to the trial;
5. Patients with significant renal function impairment (Creatinine>2mg/dl) and liver function impairment (AST and ALT > 2 x the upper limit of normal range);
6. Patients have laboratory test abnormality, which in the investigator's opinion might confound the study;
7. Patients have severe cardiac disease, e.g. unstable angina pectoris, myocardial infarction, congestive heart failure (New York Heart Association Functional Classification III and IV);
8. Patients have life threatening disease;
9. Patients are allergic to any of the composition of Chinese medicine;
10. Significant concomitant disease or medical history that could interfere with the study as judged by the investigator;

Ages: 45 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Huey-Herng Sheu, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan